CLINICAL TRIAL: NCT06236074
Title: Comparison of Modified Post-Anesthetic Discharge Scoring System (PADSS) Between 4 and 24 Hours in Patients Undergoing Laparoscopic Cholecystectomy
Brief Title: Comparison of Modified PADSS Between 4 and 24 Hours in Patients Undergoing LC
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Thammasat University Hospital (Other)
Responsible Party: Principal Investigator, Niruji Saengsomsuan, Anesthesiology, Thammasat University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: MTU-EC-AN-1-072/66
Record Dates: First submitted 2024-01-24; First posted 2024-02-01 (Actual); Last update posted 2025-09-09 (Actual); Status verified 2025-05

CONDITIONS: Laparoscopic Cholecystectomy
MeSH Terms: interventions — Cholecystectomy, Laparoscopic

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Modified Post-Anesthetic Discharge Scoring System (PADSS) between 4 and 24 hours (Other)
  Interventions: Other: Modified Post-Anesthetic Discharge Scoring System (PADSS) between 4 and 24 hours; Procedure: Laparoscopic Cholecystectomy

INTERVENTIONS:
Other: Modified Post-Anesthetic Discharge Scoring System (PADSS) between 4 and 24 hours — Observation Modified Post-Anesthetic Discharge Scoring System (PADSS) between 4 and 24 hours
Procedure: Laparoscopic Cholecystectomy — Laparoscopic Cholecystectomy

SUMMARY:
This study is compare of Modified Post-Anesthetic Discharge Scoring System (PADSS) between 4 and 24 hours in patients undergoing laparoscopic cholecystectomy

ELIGIBILITY:
Inclusion Criteria:

* Patient undergoing laparoscopic cholecystectomy
* 20-60 years old
* American Society of. Anesthesiologist physical status classification I-III

Exclusion Criteria:

* Turn to open cholecystectomy

Ages: 20 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 60 (Actual)
Dates: Start 2023-06-01 (Actual); Primary Completion 2023-12-31 (Actual); Study Completion 2025-04-30 (Actual)

PRIMARY OUTCOMES:
Comparison of Modified Post-Anesthetic Discharge Scoring System (PADSS) Between 4 and 24 Hours in Patients Undergoing Laparoscopic Cholecystectomy | 4 vs 24 hours
  The modified post-anesthetic discharge scoring system, which consists of five components (each component having 2 points): vital signs, ambulation, nausea or vomiting, pain, and surgical bleeding

CONTACTS AND LOCATIONS:
Locations (1):
- Thammasat University hospital, Pathum Thani, Klongluang, Thailand